CLINICAL TRIAL: NCT06466161
Title: Evaluation of the Agreement Between Conical Forearm and Cylindrical Upper Arm Non-Invasive Blood Pressure (NIBP) Measurements in Pregnant Patients
Brief Title: Conical Forearm and Cylindrical Upper Arm Non-Invasive Blood Pressure (NIBP) Measurements in Pregnant Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Adithya Bhat, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU00221793
Record Dates: First submitted 2024-05-31; First posted 2024-06-20 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Hypertension in Pregnancy; Hypertension; Obesity
Keywords: Hypertension; Conical Blood Pressure Cuff; Cylindrical Blood Pressure Cuff; Pregnancy; Obesity; Non invasive blood pressure
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, non blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 Upper arm cylindrical cuff (Active Comparator): In Group 1 the upper arm cylindrical cuff is inflated first and the blood pressure is measured.
  After one minute has elapsed, the forearm conical cuff is inflated and blood pressure measured.
  Interventions: Device: Upper Arm Cylindrical Blood Pressure Cuff
- Group 2 Forearm conical cuff (Experimental): In Group 2 the forearm conical cuff is inflated first and the blood pressure is measured. After one minute has elapsed, the upper arm cylindrical cuff is inflated and blood pressure measured.
  Interventions: Device: Forearm Conical Blood Pressure Cuff

INTERVENTIONS:
Device: Upper Arm Cylindrical Blood Pressure Cuff — In Group 1, the upper arm cylindrical cuff is inflated first, followed by inflation of the forearm conical cuff.
  Other Names: Upper Arm Cylindrical Blood Pressure Cuff Inflated First
  Arms: Group 1 Upper arm cylindrical cuff
Device: Forearm Conical Blood Pressure Cuff — In Group 2, the forearm conical cuff is inflated first, followed by inflation of the upper arm cylindrical cuff.
  Other Names: Forearm Conical Blood Pressure Cuff Inflated First
  Arms: Group 2 Forearm conical cuff

SUMMARY:
The diagnosis of hypertensive disease during pregnancy is predicated on strict blood pressure thresholds: 140/90 on at least two occasions measured four hours apart for both gestational hypertension and preeclampsia. An improvement in diagnostic accuracy of even 5mm Hg would be significant, as reflected by the US Association for the Advancement of Medical Instrumentation (AAMI), the British Hypertension Society, the European Society of Hypertension (ESH) Working Group on Blood Pressure (BP) Monitoring, and the International Organization for Standardization (ISO)consensus for validation of non-invasive blood pressure (NIBP) devices during pregnancy. Given the known inaccuracies of upper arm cylindrical cuff measurements in morbidly obese patients, a conical cuff which provides more accurate measurements will translate into direct patient benefit via more informed diagnosis and management. Fewer women may be exposed to unnecessary treatment, preterm delivery, and/or cesarean section. Recognizing the increasing prevalence of morbid obesity and hypertensive disease amongst pregnant women in the United States, the identification of a more accurate non-invasive cuff is desperately needed. Increasing the accuracy of NIBP measurements on Labor and Delivery has the potential to directly impact the management of tens of thousands of morbidly obese pregnant women diagnosed with hypertensive disease in the United States every year. Establishing the level of agreement between conical forearm and cylindrical upper arm cuffs will shed light on the presence and magnitude of any disparity between measurement methods.

STUDY ENDPOINTS:

Primary Outcome Measures:

* Agreement between conical and cylindrical cuff systolic blood pressure across groups
* Agreement between conical and cylindrical cuff diastolic blood pressure across groups

Secondary Outcome Measures:

• Agreement between conical and cylindrical cuff mean arterial pressure

DETAILED DESCRIPTION:
After participants have provided written informed consent they will be enrolled into one of four groups: (1) normotensive/non-obese (2) normotensive/obese (3) hypertensive/non-obese and (4) hypertensive/obese. The threshold for hypertension will be a BP measurement greater than 140/90 mmHg on two occasions at least 4 hours apart. After informed consent has been obtained, body weight (kg) and height (cm) will be measured on calibrated scales and BMI calculated. Arm circumference will be measured proximally just beneath the axilla, at mid- point between the acromion and the olecranon, and distally just above the antecubital fossa in centimeters. Forearm circumference will be measured, in millimeters, proximally just beneath the olecranon, at mid-point between the olecranon and the styloid apophysis, and distally just above the styloid apophysis. Upper arm length will be measured from the acromion to the olecranon in centimeters. Forearm length will be measured from the olecranon to the styloid apophysis in centimeters. Upper arm cuffs will be placed at the mid-point between the acromion and the olecranon processes. All BP measurements will be obtained from the participants while in the sitting position, and the arm contralateral to the peripheral intravenous catheter (PIV) will be chosen for measurement. If the PIV has not yet been placed, the arm selection will be made by the patient. Baseline BP measurement will be performed at the upper arm after at least a 5-minute resting period utilizing a large-sized cylindrical cuff. Baseline BP measurement at the forearm will be performed using a conical forearm cuff previously validated in non-pregnant patients with arm circumferences greater than or equal to 40 cm23 (RADIAL-CUF, GE HealthCare, Milwaukee, Wisconsin). The forearm cuff will be placed 3 cm from the styloid process of the ulna palpable at the wrist.

After two minutes have elapsed since the baseline measurements, sequential, paired BP measurements will then be obtained by cycling either the upper arm cylindrical cuff or forearm conical cuff, waiting 60 seconds after the measurement, then cycling the other cuff. The choice of cuff to be cycled first (conical or cylindrical) will be block randomized. Additional sequential measurements will then be obtained 2, 4, 6, 8, and 10 minutes after the first set. After the initial measurements, the upper arm cuff will automatically cycle every 15 minutes. Thus, all patients will have six sets of sequential BP measurements. Any decision to initiate antihypertensive therapy will be made by the patient's obstetrical provider, using an institutional algorithm and with reference to cylindrical cuff pressures.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18 years of age or older with a
* Body mass index (BMI) of 20 kg/m2 or greater
* Present to Labor and Delivery with or without a diagnosis of gestational hypertension, preeclampsia, or chronic hypertension with super-imposed preeclampsia, in spontaneous labor or for induction of labor

Exclusion Criteria:

* Significant peripheral arterial disease resulting in at least a 10 mm Hg blood pressure difference between both arms
* History of repaired or unrepaired congenital heart disease
* History of significant arrythmia
* History of pacemaker or implantable cardioverter defibrillator placement
* History of sickle cell disease
* History of Raynaud's phenomenon on any extremity
* History of lymph node dissection of either upper extremity
* Patients who are less than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women 18 years and older who are pregnant
Enrollment: 110 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Agreement between conical and cylindrical cuff systolic blood pressure as measured by mean absolute deviance | Through study completion, an average of 1 year
  Agreement between conical and cylindrical cuff systolic blood pressure across 4 distinct subject groups:(1) normotensive/non-obese (2) normotensive/obese (3) hypertensive/non-obese and (4) hypertensive/obese.
Agreement between conical and cylindrical cuff diastolic blood pressure as measured by mean absolute deviance | Through study completion, an average of 1 year
  Agreement between conical and cylindrical cuff diastolic blood pressure across 4 distinct groups: (1) normotensive/non-obese (2) normotensive/obese (3) hypertensive/non-obese and (4) hypertensive/obese.

SECONDARY OUTCOMES:
Agreement between conical and cylindrical cuff mean arterial pressure as measured by mean absolute deviance | Through study completion, an average of 1 year
  Agreement between conical and cylindrical cuff MAP arterial pressure among the 4 distinct groups:(1) normotensive/non-obese (2) normotensive/obese (3) hypertensive/non-obese and (4) hypertensive/obese.
Likert scale patient satisfaction scores for conical and cylindrical cuff measurements | Through study completion, an average of 1 year
  Patient satisfaction scores for conical and cylindrical cuff measurements will be measured with a 5-question survey using 5-point scale, ranging from 0 (very painful/very dissatisfied) to 5 (not painful at all/very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Adithya Bhat, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists. ACOG Committee opinion no. 549: obesity in pregnancy. Obstet Gynecol. 2013 Jan;121(1):213-7. doi: 10.1097/01.aog.0000425667.10377.60. PMID 23262963
- [Background] Crane JM, Murphy P, Burrage L, Hutchens D. Maternal and perinatal outcomes of extreme obesity in pregnancy. J Obstet Gynaecol Can. 2013 Jul;35(7):606-611. doi: 10.1016/S1701-2163(15)30879-3. PMID 23876637
- [Background] Chu SY, Kim SY, Lau J, Schmid CH, Dietz PM, Callaghan WM, Curtis KM. Maternal obesity and risk of stillbirth: a metaanalysis. Am J Obstet Gynecol. 2007 Sep;197(3):223-8. doi: 10.1016/j.ajog.2007.03.027. PMID 17826400
- [Background] Lutsiv O, Mah J, Beyene J, McDonald SD. The effects of morbid obesity on maternal and neonatal health outcomes: a systematic review and meta-analyses. Obes Rev. 2015 Jul;16(7):531-46. doi: 10.1111/obr.12283. Epub 2015 Apr 24. PMID 25912896
- [Background] Bicocca MJ, Mendez-Figueroa H, Chauhan SP, Sibai BM. Maternal Obesity and the Risk of Early-Onset and Late-Onset Hypertensive Disorders of Pregnancy. Obstet Gynecol. 2020 Jul;136(1):118-127. doi: 10.1097/AOG.0000000000003901. PMID 32541276
- [Background] Bodnar LM, Catov JM, Klebanoff MA, Ness RB, Roberts JM. Prepregnancy body mass index and the occurrence of severe hypertensive disorders of pregnancy. Epidemiology. 2007 Mar;18(2):234-9. doi: 10.1097/01.ede.0000254119.99660.e7. PMID 17237733
- [Background] O'Brien TE, Ray JG, Chan WS. Maternal body mass index and the risk of preeclampsia: a systematic overview. Epidemiology. 2003 May;14(3):368-74. doi: 10.1097/00001648-200305000-00020. PMID 12859040
- [Background] Lisonkova S, Joseph KS. Incidence of preeclampsia: risk factors and outcomes associated with early- versus late-onset disease. Am J Obstet Gynecol. 2013 Dec;209(6):544.e1-544.e12. doi: 10.1016/j.ajog.2013.08.019. Epub 2013 Aug 22. PMID 23973398
- [Background] Lisonkova S, Sabr Y, Mayer C, Young C, Skoll A, Joseph KS. Maternal morbidity associated with early-onset and late-onset preeclampsia. Obstet Gynecol. 2014 Oct;124(4):771-781. doi: 10.1097/AOG.0000000000000472. PMID 25198279
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] Creanga AA, Syverson C, Seed K, Callaghan WM. Pregnancy-Related Mortality in the United States, 2011-2013. Obstet Gynecol. 2017 Aug;130(2):366-373. doi: 10.1097/AOG.0000000000002114. PMID 28697109
- [Background] Cantwell R, Clutton-Brock T, Cooper G, Dawson A, Drife J, Garrod D, Harper A, Hulbert D, Lucas S, McClure J, Millward-Sadler H, Neilson J, Nelson-Piercy C, Norman J, O'Herlihy C, Oates M, Shakespeare J, de Swiet M, Williamson C, Beale V, Knight M, Lennox C, Miller A, Parmar D, Rogers J, Springett A. Saving Mothers' Lives: Reviewing maternal deaths to make motherhood safer: 2006-2008. The Eighth Report of the Confidential Enquiries into Maternal Deaths in the United Kingdom. BJOG. 2011 Mar;118(Suppl 1):1-203. doi: 10.1111/j.1471-0528.2010.02847.x. PMID 21356004
- [Background] Babbs CF. Oscillometric measurement of systolic and diastolic blood pressures validated in a physiologic mathematical model. Biomed Eng Online. 2012 Aug 22;11:56. doi: 10.1186/1475-925X-11-56. PMID 22913792
- [Background] Mauck GW, Smith CR, Geddes LA, Bourland JD. The meaning of the point of maximum oscillations in cuff pressure in the indirect measurement of blood pressure--part ii. J Biomech Eng. 1980 Feb;102(1):28-33. doi: 10.1115/1.3138195. PMID 7382450
- [Background] Palatini P, Benetti E, Fania C, Malipiero G, Saladini F. Rectangular cuffs may overestimate blood pressure in individuals with large conical arms. J Hypertens. 2012 Mar;30(3):530-6. doi: 10.1097/HJH.0b013e32834f98a0. PMID 22278143
- [Background] Palatini P, Parati G. Blood pressure measurement in very obese patients: a challenging problem. J Hypertens. 2011 Mar;29(3):425-9. doi: 10.1097/HJH.0b013e3283435b65. No abstract available. PMID 21317721
- [Background] Kho CL, Brown MA, Ong SL, Mangos GJ. Blood pressure measurement in pregnancy: the effect of arm circumference and sphygmomanometer cuff size. Obstet Med. 2009 Sep;2(3):116-20. doi: 10.1258/om.2009.090017. Epub 2009 Sep 1. PMID 27582825
- [Background] Schoenfeld A, Ziv I, Tzeel A, Ovadia J. Roll-over test--errors in interpretation, due to inaccurate blood pressure measurements. Eur J Obstet Gynecol Reprod Biol. 1985 Jan;19(1):23-30. doi: 10.1016/0028-2243(85)90161-3. PMID 3979651
- [Background] Stergiou GS, Alpert B, Mieke S, Asmar R, Atkins N, Eckert S, Frick G, Friedman B, Grassl T, Ichikawa T, Ioannidis JP, Lacy P, McManus R, Murray A, Myers M, Palatini P, Parati G, Quinn D, Sarkis J, Shennan A, Usuda T, Wang J, Wu CO, O'Brien E. A Universal Standard for the Validation of Blood Pressure Measuring Devices: Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO) Collaboration Statement. Hypertension. 2018 Mar;71(3):368-374. doi: 10.1161/HYPERTENSIONAHA.117.10237. Epub 2018 Jan 31. PMID 29386350
- [Background] Palatini P, Asmar R. Cuff challenges in blood pressure measurement. J Clin Hypertens (Greenwich). 2018 Jul;20(7):1100-1103. doi: 10.1111/jch.13301. PMID 30003699
- [Background] Leblanc ME, Croteau S, Ferland A, Bussieres J, Cloutier L, Hould FS, Biertho L, Moustarah F, Marceau S, Poirier P. Blood pressure assessment in severe obesity: validation of a forearm approach. Obesity (Silver Spring). 2013 Dec;21(12):E533-41. doi: 10.1002/oby.20458. Epub 2013 Jun 22. PMID 23512945
- [Background] Leblanc ME, Auclair A, Leclerc J, Bussieres J, Agharazii M, Hould FS, Marceau S, Brassard P, Godbout C, Grenier A, Cloutier L, Poirier P. Blood Pressure Measurement in Severely Obese Patients: Validation of the Forearm Approach in Different Arm Positions. Am J Hypertens. 2019 Jan 15;32(2):175-185. doi: 10.1093/ajh/hpy152. PMID 30312368
- [Background] Hersh LT, Sesing JC, Luczyk WJ, Friedman BA, Zhou S, Batchelder PB. Validation of a conical cuff on the forearm for estimating radial artery blood pressure. Blood Press Monit. 2014 Feb;19(1):38-45. doi: 10.1097/MBP.0000000000000011. PMID 24217368
- [Background] Palatini P, Benetti E, Fania C, Saladini F. Only troncoconical cuffs can provide accurate blood pressure measurements in people with severe obesity. J Hypertens. 2019 Jan;37(1):37-41. doi: 10.1097/HJH.0000000000001823. PMID 29927843